CLINICAL TRIAL: NCT05142501
Title: Observation of Humoral and Cellular Immune Response After Additional Vaccine Dose With Different COVID-19 Vaccines in ESKD Patients in Hemodialysis Therapy
Brief Title: Observation of the Immune Response After COVID-19 Additional Vaccine Doses in Chronic Patients in Hemodialysis Therapy
Acronym: COVID-thIRd
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: HD-COVID-IR-EU
Record Dates: First submitted 2021-12-01; First posted 2021-12-02 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Chronic Kidney Diseases; COVID-19; Hemodialysis
Keywords: Chronic Kidney Disease; COVID-19; Immune responses
MeSH Terms: conditions — Renal Insufficiency, Chronic; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood samples — Four consecutive blood sampling throughout the overall follow-up period of 12 months.

SUMMARY:
Observation of humoral and cellular immune response after additional dose vaccine with different COVID-19 vaccines in ESKD patients in hemodialysis therapy.

DETAILED DESCRIPTION:
In this open, prospective, observational trial the humoral and cellular immune response in ESKD patients undergoing hemodialysis shall be analyzed after administration of a fourth dose of vaccine. The total follow-up time per patient is up to 12 months after the fourth dose of vaccine.

In total, 340 patients (170 patients per country) shall be included. Only adult patients capable of giving consent will be enrolled. The humoral immune response will be analyzed in all patients, whereas the analysis of the cellular immune response will only be conducted in 15% of the enrolled patients.

The HD-COVID-IR-EU study shall be conducted in Portugal and in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by study patient and investigator/authorized physician
* Minimum age of 18 years
* Ability to understand the nature and requirements of the study
* ESKD patients on maintenance hemodialysis with a minimum of 4hrs three times a week at the time of recruitment and a dialysis vintage ≥3 months in NC clinics
* Patients that already received three doses against COVID-19 as detailed in the manufacturer's instructions
* Patients that are scheduled to receive a fourth vaccine dose of either Comirnaty (BioNTech/Pfizer) or Spikevax (Moderna) after approval of respective national authority.

Exclusion Criteria:

* Any conditions which could interfere with the patient's ability to comply with the study
* Participation in an interventional clinical study during the preceding 30 days
* Previous participation in the same study
* Patients with proven current COVID-19 infection as identified by routine clinical practice
* Patient in therapy with immunosuppressive medications / immunomodulators
* Patients who already received a fourth COVID-19 vaccination dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prevalent hemodialysis patients treated who receive three hemodialysis treatments per week.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Humoral immune response | 12 months after start of study
  The humoral immune response will be assessed at four different timepoints (Sample 1: prior to the fourth vaccine dose; sample 2: 1 months after the fourth vaccine dose; sample 3: 6 months after the fourth vaccine dose; sample 4: 12 months after the fourth vaccine dose or max. 4 weeks prior to the fifth vaccine dose, whichever comes first) through the measurement of the titers of Bioplex IgG antibody panel in study participant's blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ponce, Dr, Principal Investigator — Nephrocare Portugal; Maria Eva Baró Salvador, Dr, Principal Investigator — Fresenius Medical Care España, S.A.U.
Locations (11):
- Portugal (4):
  - NephroCare Amadora, Amadora
  - NephroCare Restelo, Lisbon
  - NephroCare Lumiar, Lisbon
  - NephroCare Vila Franca de Xira, Vila Franca de Xira
- Spain (7):
  - Centro de Diálisis Barcelona - Glories, Barcelona
  - Centro de Diálisis Barcelona - Rosselló, Barcelona
  - Centro de Diálisis Granollers, Granollers
  - Centro de Diálisis Dialcentro, Madrid
  - Centro de Diálisis San Luciano, Madrid
  - Centro de Diálisis Sant Boi, Sant Boi de Llobregat
  - Centro de Diálisis Terrassa, Terrassa

IPD SHARING:
Plan to Share IPD: No